CLINICAL TRIAL: NCT02141412
Title: Intravenous Dexmedetomidine For The Quaity Of Emergence From General Anesthesia: A Dose-Finding Study
Brief Title: Intravenous Dexmedetomidine For The Quaity Of Emergence From General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Professor of Clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANES.MA.10
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia Recovery; Anesthesia Emergence; Shivering; Postoperative Recovery
Keywords: optimal dose of dexmedetomidine; prevent shivering; improve quality of emergence; anesthesia; without delay; recovery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group I (Active Comparator): Patients in Group I will receive dexmedetomidine 0.25 µg/kg IV (over 10 min) at closure of sevoflurane
  Interventions: Drug: dexmedetomidine 0.25 µg/kg IV
- Group II (Active Comparator): Patients in Group II will receive dexmedetomidine 0.5 µg/kg IV (over 10 min) at closure of sevoflurane
  Interventions: Drug: dexmedetomidine 0.5 µg/kg IV
- Group III (Active Comparator): Patients in Group III will receive dexmedetomidine 1 µg/kg IV (over 10 min) at closure of sevoflurane
  Interventions: Drug: dexmedetomidine 1 µg/kg IV
- Group IV (Placebo Comparator): Patients in Group IV will receive same volume of normal saline at closure of sevoflurane
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: dexmedetomidine 0.25 µg/kg IV
  Arms: Group I
Drug: dexmedetomidine 0.5 µg/kg IV
  Arms: Group II
Drug: dexmedetomidine 1 µg/kg IV
  Arms: Group III
Drug: Placebo Comparator — Patients in Group IV will receive same volume of normal saline at closure of sevoflurane
  Arms: Group IV

SUMMARY:
In a prospective randomized clinical trial involving adult patients undergoing elective surgery under general anesthesia, the investigators will enroll 216 patients, and evaluate 3 doses of prophylactic dexmedetomidine as a means to reduce postoperative shivering and quality of emergence from anesthesia versus placebo.

DETAILED DESCRIPTION:
Patients undergoing surgery under general anesthesia may experience several complications during the postoperative period. Shivering has been reported to occur in up to 65% of patients recovering from general anesthesia, and has been shown to cause detrimental effects to the patient. Previous studies have shown that dexmedetomidine 1µg/kg at the end of surgery significantly reduces the incidence of postoperative shivering and improves quality of emergence from anesthesia. However, this beneficial effect of dexmedetomidine is at the expense of prolonged time to extubation and awakening. The aim of this study is to find the optimal dose of dexmedetomidine that would be beneficial without delaying recovery from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year-old
* ASA class I, II, and III
* patients undergoing elective surgery under general anesthesia with an estimated time of 1-3 h

Exclusion Criteria:

* duration of surgery less than 1h or more than 3 h
* allergy to dexmedetomidine
* vasoactive antidepressant or analgesics
* obesity (BMI>30)
* fever
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postanaesthetic shivering incidence and score | change from baseline every 10 minutes up to 1 hour post-operatively
Quality of emergence from anesthesia | Change from baseline every 5 minutes till extubation
  The anesthesiologist blinded to the group allocation will assess patients for coughing, hypertension, tachycardia, limb movement during extubation

SECONDARY OUTCOMES:
Patient's Temperature | every 10 minutes up to 1 hour post-operatively
Time to extubation, awakening and orientation | 1 hour post-operatively
Sedation scores | every 10 minutes up to 1 hour post-operatively
Pain scores | every 10 minutes up to 1 hour post-operatively
Nausea and vomiting | every 10 minutes up to 1 hour post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Marie Aouad, MD, Principal Investigator — American Univesity of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon